CLINICAL TRIAL: NCT04904718
Title: Real World Evaluation of Advisor Pro in Clinical Practice
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Decided not to proceed with enrollment - study never started
Sponsor: Yale University (Other)
Collaborators: DreaMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2000029019
Record Dates: First submitted 2021-05-19; First posted 2021-05-27 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Type1diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DreaMed Advisor Pro tool used for insulin optimization (Experimental)
  Interventions: Device: DreaMed Advisor Pro

INTERVENTIONS:
Device: DreaMed Advisor Pro — Advisor Pro software is a proprietary algorithm, designed to provide a comprehensive analysis of individual diabetes data consisting of glucose levels, insulin delivery history and meal consumption reported

SUMMARY:
To assess the integration of the DreaMed Advisor Pro tool into a real-world clinical practice using both in person and virtual visits to assess benefits in glycemia, as measured by the glucose management indicator and other glucose metrics.

To determine acceptability of the DreaMed Advisor Pro tool both from a person with diabetes as well as a health care provider perspective.

To quantify the potential reimbursement potential that could be generated with use of the DreaMed Advisor Pro.

ELIGIBILITY:
Inclusion Criteria:

1. Participant with Type 1 diabetes
2. Age ≥ 6 years to <30 years
3. Using Insulin infusion pump (CSII) therapy including those with low glucose suspend and predictive low glucose suspend features

   1. Insulin pump must not use automated insulin delivery (closed loop, artificial pancreas)
   2. Total daily dose of insulin must be greater than 0.5 units/kg/day
4. Participants / parents are required to have minimum computer skills and access to a computer in order to upload their personal devices (Pump, BG meter etc) to Tidepool.
5. Participants using Dexcom sensors will allow access to their account for the study duration
6. Participants not using CGM must agree to test BG at least 4 times a day at appropriate intervals
7. Participants / parents will have to have a smartphone (Apple or Android and Windows)

Exclusion Criteria:

1. An episode of diabetic ketoacidosis within the month prior to study entry
2. Any significant diseases / conditions including psychiatric disorders and substance abuse that in the opinion of the investigator is likely to affect the subject's ability to complete the study or compromise patient's safety,
3. Current participation in any other interventional study
4. Female subject who is pregnant or lactating or planning to become pregnant within the planned study duration
5. Severe hypoglycemia within six months prior to enrollment as defined by the ADA and Endocrine Society
6. Current use of the following medications: medications that are used to lower blood glucose such as Pramlintide, Metformin and GLP-1 analogs. Beta blockers, glucocorticoids and other medications, which in the judgment of the investigator would be a contraindication to participation in the study (Anticoagulant therapy e.g. Plavix, LMW heparin, Coumadin, Immunosuppressant therapy)
7. Participants suffers from an eating disorder

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in glucose control with the use of DreaMed | 6 months
  Glucose mangement indicator (GMI) will be used to determine glucose control. The GMI indicates the average A1C level that would be expected based on mean glucose measured in a large number of individuals with diabetes. Mean glucose ideally is derived from at least 14 days of CGM data

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Sherr, MD, PhD, Principal Investigator — Yale University

IPD SHARING:
Plan to Share IPD: No